CLINICAL TRIAL: NCT02184377
Title: The Function of Cricothyroid Muscle and Its Impaction on Mandarin Lexical Tones in Unilateral Vocal Fold Paralysis: a Quantified Laryngeal Electromyography Based Research
Brief Title: The Function of Cricothyroid Muscle and Its Impaction on Mandarin Lexical Tones in Unilateral Vocal Fold Paralysis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Fang Tuan-Jen, Director, Laryngology, Chang Gung Memorial Hospital
Other Study IDs: 101_4920A3
Record Dates: First submitted 2014-06-23; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Unilateral Vocal Cord Paralysis
Keywords: quantitative laryngeal electromyography; cricothyroid muscle; unilateral vocal fold paralysis; superior laryngeal nerve; lexical tone; Mandarin
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RLN+SLN paralysis: unilateral recurrent laryngeal and superior laryngeal nerve paralysis
- RLN paralysis: unilateral recurrent laryngeal nerve paralysis

SUMMARY:
Mandarin Chinese phonemically distinguishes four tones, with Tone 1 having high-level pitch, Tone 2 high-rising pitch, Tone 3 low-dipping pitch, and Tone 4 high-falling pitch The same segmental context carries different meanings depending on the tone. The function deficit of cricothyroid (CT) muscle, innervated by external branch superior laryngeal nerve (eSLN), would impair the speech tone adjustment. The defect in tone adjustment may interfere with the communication function in Mandarin Chinese speaker more than other language users. This may explain while peripheral unilateral vocal fold paralysis (UVFP) patients with eSLN injury had worse outcomes than those with sole recurrent laryngeal nerve paralysis. The neuromuscular control of laryngeal muscle can be evaluated by laryngeal electromyography (LEMG). The investigators have utilized a quantified LEMG (denoted Q-LEMG) in their previous research to measure the neuromuscular control of thyroarytenoid- lateral cricoarytenoid (TA-LCA) adductor complex. However, the task to measure the CT muscle function by Q-LEMG has not been developed yet. It is of thus of utmost interest to develop a standardized task to measure the neuromuscular function of CT muscle in Mandarin speakers. In Mandarin speaking patients with UVFP, the lexical tone influence from CT muscle can be discovered by the technique. The investigators also want to measure the lexical tone correction by conventional laryngoplasty and its influence in CT muscle activity. The data of lexical tone and its correlation with CT contractile activity is important in attempting pitch adjust artificial electrolarynx.

DETAILED DESCRIPTION:
Purposes: 1. Searching for a standard task to measure CT function by Q-LEMG. 2. Correlate the data among Q-LEMG activity of CT muscle, lexical tone in Mandarin and vocal cord position and its impaction on vocal functions. 3. Detect the influence of lexical tone from conventional laryngoplasty for peripheral UVFP with eSLN injury.

Study designs: The current research is a two-year study. In the first year, the investigators will develop a standardized task for quantified LEMG analysis for CT muscles which were controlled by eSLN. In the second year, patients with acute UVFP will be enrolled into the study. By comprehensive evaluation including Q-LEMG analysis, the impact of injection laryngoplasty on tone adjustment can be identified. The results between UVFP with or without CT muscle damage will also be compared.

Predictive outcomes: 1. Developing a standard tool, Q-LEMG, to measure the function CT muscles. 2. Achieve the correlation of the neuromuscular control of lexical tone and CT muscle. 3. Analyze the impaction of early temporary injection on speech modal tone in Mandarin speakers and neuromuscular control in CT muscles. 4. Applying the data of tone and CT signals to future pitch controlled artificial electrolarynx animal models.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute unilateral vocal palsy
* Patients with clear conscious and stable mental status

Exclusion Criteria:

* Patients with wounds on the neck or with bleeding disorder or serious cardiopulmonary dysfunction
* Patients who cannot sit for longer than 30 minutes or received other vocal cord treatments before the selection
* Pregnant and breastfeeding women
* Patients with communication disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a tertian referral medical center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
laryngeal electromyography | before hyaluronate injection; one month after hyaluronate injection

SECONDARY OUTCOMES:
laboratory voice analysis | before hyaluronate injection; one month after hyaluronate injection
  The voice analysis:
  fundamental frequency, Jitter (perturbation of frequency), Shimmer (perturbation of amplitude), harmonic-to-noise ratio (HN), and s/z ratio (SZ) .
voice outcomes survey (VOS) | before hyaluronate injection; one month after hyaluronate injection
  questionnaire
Short form -36 | before hyaluronate injection; one month after hyaluronate injection
  questionnaire
voice range profile | before hyaluronate injection; one month after hyaluronate injection
  The voice will be analyzed by computerized software. The extreme lowest and highest notes of frequencies production and the amplitude will be recorded and a voice map will be made as a plot of sound pressure level versus F0.

CONTACTS AND LOCATIONS:
Overall Officials: Tuan-Jen Fang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkuo, Taiwan